CLINICAL TRIAL: NCT02148120
Title: A Phase II, Multicentre, Double-blind, Randomised, 5-way Crossover Study to Test the Non-inferiority of the Acute Bronchodilator Effect of CHF 1535 200/6 µg NEXThaler Versus CHF 1535 100/6 µg NEXThaler in Partially Controlled and Uncontrolled Adult Asthmatic Patients.
Brief Title: A Study to Evaluate the Acute Bronchodilator Effect of CHF1535 NEXThaler
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-01535BA1-01
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CHF1535 NEXThaler 100/6, 1 puff (Active Comparator): Beclometasone Dipropionate 100 µg + Formoterol Fumarate 6 µg
  Interventions: Drug: Beclometasone Dipropionate 100 µg + Formoterol Fumarate 6 µg
- CHF1535 NEXThaler 100/6 µg, 4 puffs (Active Comparator): Beclometasone Dipropionate 400 µg + Formoterol Fumarate 24 µg
  Interventions: Drug: Beclometasone Dipropionate 100 µg + Formoterol Fumarate 6 µg
- CHF1535 NEXThaler 200/6 µg, 1 puff (Experimental): Beclometasone Dipropionate 200 µg + Formoterol Fumarate 6 µg
  Interventions: Drug: Beclometasone Dipropionate 200 µg + Formoterol Fumarate 6 µg
- CHF1535 NEXThaler 200/6 µg, 4 puffs (Experimental): Beclometasone Dipropionate 800 µg + Formoterol Fumarate 24 µg
  Interventions: Drug: Beclometasone Dipropionate 200 µg + Formoterol Fumarate 6 µg
- Placebo NEXThaler (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beclometasone Dipropionate 100 µg + Formoterol Fumarate 6 µg
  Other Names: Foster NEXThaler
  Arms: CHF1535 NEXThaler 100/6 µg, 4 puffs; CHF1535 NEXThaler 100/6, 1 puff
Drug: Beclometasone Dipropionate 200 µg + Formoterol Fumarate 6 µg
  Arms: CHF1535 NEXThaler 200/6 µg, 1 puff; CHF1535 NEXThaler 200/6 µg, 4 puffs
Drug: Placebo
  Arms: Placebo NEXThaler

SUMMARY:
The aim of the study is to demonstrate the non-inferiority in terms of acute bronchodilator effect between a single dose of CHF 1535 NEXThaler 200/6 µg and a single dose of CHF 1535 NEXThaler 100/6 µg at two dose levels in partially controlled and uncontrolled asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written informed consent obtained prior to any study-related procedures.
* Male or female aged between 18 and 65 years inclusive;
* Evidence for "partially controlled" or "uncontrolled" asthma;
* Medium daily dose of previous inhaled corticosteroids (ICS) treatment;
* FEV1 between 60% and 85% of the predicted normal values;
* A documented positive response to the reversibility test;
* Non-smokers or ex-smokers;
* A cooperative attitude and ability to be trained in the proper use of a DPI.

Exclusion Criteria:

* Pregnant or lactating women and all women physiologically capable of becoming pregnant not willing to use at least one acceptable method of contraception.
* Significant seasonal variation in asthma occurring or expected to occur during study participation;
* History of near fatal asthma, brittle asthma, accident and Emergency treatment or hospitalisation for asthma exacerbation in Intensive Care Unit within 1 year before screening;
* Occurrence of asthma exacerbations or respiratory tract infections in the 4 weeks preceding the screening;
* Diagnosis of Chronic Obstructive Pulmonary Disease;
* History of cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency;
* Diagnosis of restrictive lung disease;
* Patients treated with oral or parenteral corticosteroids in the previous 8 weeks;
* Intolerance or contra-indication to treatment with beta2-agonists and/or inhaled corticosteroids;
* Allergy, sensitivity or intolerance to study drugs or excipients;
* Patients who received any investigational drug within the last 8 weeks before the screening;
* Patients taking any of the non-permitted concomitant medication;
* Subjects unlikely to comply with the study protocol;
* Any clinically relevant abnormal value or physical finding at screening;
* Significant medical history;
* Abnormal and clinically significant 12-lead electrocardiogram;
* Patients with low compliance of QVAR intake.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
FEV1 Area under the curve | until 12 h post dose
  FEV1= Forced expiratory volume in the first second of expiration

SECONDARY OUTCOMES:
FEV1 peak | until 12 h post dose
  Maximum FEV1 value
FVC area under the curve | until 12 h post dose
  FVC = Forced Vital Capacity
FVC peak | until 12 h post dose
  Maximum FVC
Adverse events | over a period of 5 to 14 weeks
  from the signature of the informed consent until the end of the study, the total duration depends on the duration of the run-in and wash-out periods.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Hammersmith Medicines Research, London
  - Respiratory Clinical Trials, Hearth Lung Centre, London
  - Medicines Evaluation Unit, Manchester

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2013-004826-27